CLINICAL TRIAL: NCT05511415
Title: In Vitro Evaluation of Spontaneous and Oxytocin-induced Contractility of Pregnant Human Myometrium During Exposure to Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-05
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-01

CONDITIONS: Postpartum Hemorrhage
Keywords: uterine contraction; oxytocin; dexmedetomidine
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dexmedetomidine (Active Comparator): The myometrial samples are bathed in increasing concentrations of dexmedetomidine (from 10 -9M to 10 -4M).
  Interventions: Drug: Dexmedetomidine
- Oxytocin (Active Comparator): The myometrial samples are bathed in oxytocin 20nM.
  Interventions: Drug: Oxytocin
- Dexmedetomidine + Oxytocin (Active Comparator): The myometrial samples are bathed in oxytocin at 20nM along with dexmedetomidine (10-9M to 10-4M).
  Interventions: Drug: Oxytocin; Drug: Dexmedetomidine
- Oxytocin pre-treatment followed by Dexmedetomidine (Active Comparator): The myometrial samples are pre-treated with oxytocin (10-5M) for 2 hours, and then in increasing concentrations of dexmedetomidine (from 10 -9M to 10 -4M).
  Interventions: Drug: Oxytocin; Drug: Dexmedetomidine
- Oxytocin pre-treatment followed by Oxytocin (Active Comparator): The myometrial samples are pre-treated with oxytocin (10-5M) for 2 hours, and then bathed in oxytocin at 20nM.
  Interventions: Drug: Oxytocin
- Oxytocin pre-treatment followed by Dexmedetomidine + Oxytocin (Active Comparator): The myometrial samples are pre-treated with oxytocin (10-5M) for 2 hours, and then bathed in oxytocin at 20nM along with dexmedetomidine (10-9M to 10-4M)
  Interventions: Drug: Oxytocin; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Oxytocin — Oxytocin solution, 20nM concentration
  Other Names: pitocin
  Arms: Dexmedetomidine + Oxytocin; Oxytocin; Oxytocin pre-treatment followed by Dexmedetomidine; Oxytocin pre-treatment followed by Dexmedetomidine + Oxytocin; Oxytocin pre-treatment followed by Oxytocin
Drug: Dexmedetomidine — Dexmedetomidine (10-9M to 10-4M)
  Arms: Dexmedetomidine; Dexmedetomidine + Oxytocin; Oxytocin pre-treatment followed by Dexmedetomidine; Oxytocin pre-treatment followed by Dexmedetomidine + Oxytocin

SUMMARY:
Postpartum hemorrhage (PPH) remains to be one of the leading causes of maternal morbidity and mortality. It has been noted that an increasing number of PPH is attributed to the increased incidence of uterine atony. Myometrial contraction is affected by the choice of anesthetic technique and medications during cesarean delivery (CD). It has been proven that exposure to oxytocin during labor results in a decrease in myometrial contractions.

Dexmedetomidine is a drug which has been used in obstetric practice due to its desirable effects such as decreasing pain, reduced elevation in blood pressure and heart rate, sedation, and diminished anesthetic requirement. It has been used as an adjunct during spinal or epidural anesthesia during CD and even during general anesthesia for some obstetric surgeries.

The use of dexmedetomidine has been continuously rising due to its favorable effects. Its use as an adjunct in general anesthesia for obstetrical surgeries has been shown to have promising advantages. During this pandemic, dexmedetomidine has been utilized largely as a sedative in critically ill and intubated patients. This does not exclude critically ill pregnant patients who may also need to deliver urgently. Thus, it is important to investigate its effect on uterine contractility on this particular group of patients.

The investigators hypothesize that dexmedetomidine causes a dose-dependent increase in contractility of the pregnant human myometrium, both spontaneous and oxytocin-induced.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients scheduled for elective CD under regional anesthesia at 37-41 weeks of gestational age will be included in this study.
* Only patients for primary CD or repeat CD (1x) will be included in this study since excessive uterine scarring from multiple CD may affect the contractility of myometrial sample.

Exclusion Criteria:

* patient refusal
* emergency CD
* general anesthesia
* placenta accreta spectrum disorder
* any condition predisposing the patient to uterine atony (e.g. polyhydramnios, multiple gestation)
* patients taking medications affecting myometrial contractions(labetalol, magnesium etc.).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Motility index | 4 hours
  Motility index (MI) is a calculated outcome, based on the formula: frequency/(10 x amplitude).
  Frequency and amplitude are secondary outcome measures as described below.
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.

SECONDARY OUTCOMES:
Amplitude of contraction | 4 hours
  The maximum extent of uterine muscle contraction, measured in grams (g). The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Frequency of contraction | 4 hours
  The number of contractions in uterine muscle (myometrium) over 10 minutes, spontaneously and in response to an agonist. The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Integrated area under response curve (AUC) | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No